CLINICAL TRIAL: NCT00995722
Title: Efficacy of Prednisone In the Treatment of Ocular Myasthenia: The EPITOME' Study
Brief Title: Efficacy of Prednisone In the Treatment of Ocular Myasthenia
Acronym: EPITOME'
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: Michael Benatar (Other)
Collaborators: University of Miami (Other); University of Rochester (Other)
Responsible Party: Sponsor-Investigator, Michael Benatar, MBChB, DPhil, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FD-R-03710-01
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Ocular Myasthenia Gravis
Keywords: Ocular myasthenia gravis; Prednisone; Steroids
MeSH Terms: conditions — Myasthenia Gravis | interventions — Prednisone; Steroids; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone + Pyridostigmine (Experimental): Corticosteroid
  Interventions: Drug: Prednisone
- Placebo + Pyridostigmine (Placebo Comparator): Matched, inactive substance
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — Prednisone will be adjusted based on combined measures of tolerability and efficacy. Capsules will contain 10mg of prednisone.
  Other Names: Steroid
  Arms: Prednisone + Pyridostigmine
Drug: Placebo — Placebo dosages will be adjusted based on combined measures of tolerability and efficacy. Capsules will contain matching placebo.
  Other Names: Sugar pill
  Arms: Placebo + Pyridostigmine

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of prednisone in patients diagnosed with ocular myasthenia.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
The purpose of this study is to learn two things about prednisone in patients with ocular myasthenia. The first thing we aim to learn is whether or not prednisone is effective in improving the symptoms of double vision and drooping eyes that are experienced by patients with ocular myasthenia. The second thing we aim to learn is whether we can find a dose of prednisone that is well tolerated and safe. The overall goal is to find out whether a dose of prednisone that is safe and well tolerated is also effective in improving the symptoms of ocular myasthenia.

After completing screening assessments to confirm eligibility, all participants will receive treatment with pyridostigmine. If a participant's symptoms do not resolve within the first month while being treated with pyridostigmine, they will be randomized to receive prednisone or placebo. The amount of study medication a participant receives will depend on how their symptoms respond to the medication and if they experience any side effects.

After four months, participants that continue to have symptoms of ocular myasthenia and do not have side effects will receive open label high dose prednisone. Participants that no longer have symptoms will taper their dose of study drug in a double-blind fashion.

ELIGIBILITY:
Inclusion Criteria:

* Weakness confined to the extra-ocular muscles, eyelid levator and eye closure with an ocular-QMG1 score ≥ 1
* At least one of the following combinations of abnormal diagnostic testing: a) Elevated acetylcholine receptor antibody titers, (b) Abnormal repetitive nerve stimulation (> 10% decrement following slow repetitive nerve stimulation) of any nerve-muscle pair, (c) Abnormal jitter on single fiber or concentric needle electromyography in any muscle, (d) Positive ice test and brain MRI that demonstrates no central nervous system pathology that mimics ocular myasthenia, or (e) Positive Tensilon test and brain MRI that demonstrate no central nervous system pathology that mimics ocular myasthenia
* Either no prior treatment with pyridostigmine, or participant has persistent ocular symptoms that are functionally limiting or troublesome despite treatment with pyridostigmine.
* Age 18 years or older, male or female
* Capable of providing informed consent and complying with study procedures
* Identifiable primary care physician to assist with management of medical complications that may arise as a consequence of steroid therapy
* Willing to be randomized to a trial of prednisone or placebo if symptoms respond inadequately to pyridostigmine.

Exclusion Criteria:

* Disease duration (time since symptom onset) > 5 years
* Treatment with prednisone or other corticosteroids within 90 days of randomization
* Treatment with azathioprine, cyclosporine, mycophenolate mofetil or other immune suppressive medication since onset of MG unless dosages of these medications and/or duration of therapy with these medications are clinically insignificant in the judgment of the PI
* Intravenous immunoglobulin or plasma exchange within 90 days of randomization
* Prior thymectomy or history of thymoma
* Contraindication to steroids (poorly controlled diabetes, glaucoma or hypertension, history of prior steroid intolerance, obesity [BMI > 39.9kg/m2] or a history of osteoporotic fracture)
* Pregnant or lactating
* Renal failure, active thyroid or hepatocellular disease, chronic infection, poorly controlled cardiac disease, unstable psychiatric illness, untreated major depression or any other illness that would, in the opinion of the treating neurologist, make it unsafe for the patient to participate in the trial
* Receipt of another investigational drug within 30 days of Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Benatar, MBChB, DPhil, Principal Investigator — University of Miami; Gil Wolfe, MD, Study Director — State University of New York at Buffalo; Donald Sanders, MD, Study Director — Duke University
Locations (10):
- United States (8):
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - University at Buffalo, Buffalo General Medical Center, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Toronto General Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisone: Corticosteroid
  Prednisone: Prednisone will be adjusted based on combined measures of tolerability and efficacy. Capsules will contain 10mg of prednisone.
  Pyridostigmine: Prior to randomization, pyridostigmine dosage increments will be made as needed for myasthenic symptoms and as tolerated according to a pre-specified dosage titration schedule. Following randomization, dose will remain constant.
- Placebo: Matched, inactive substance
  Placebo: Placebo dosages will be adjusted based on combined measures of tolerability and efficacy. Capsules will contain matching placebo.
  Pyridostigmine: Prior to randomization, pyridostigmine dosage increments will be made as needed for myasthenic symptoms and as tolerated according to a pre-specified dosage titration schedule. Following randomization, dose will remain constant.
Period: Double Blinded: 16 Weeks
Arm/Group | Prednisone | Placebo
Started | 6 | 5
Completed | 5 | 4
Not Completed | 1 | 1
Period: Overall Study: 36 Weeks
Arm/Group | Prednisone | Placebo
Started | 5 | 4
Completed | 3 | 2
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (18) | 62 (9) | 63 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: Failure to achive sustatined minimal manifestation status by week 16
Time Frame: 4 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 5
percentage of participants | 17 [0 to 64] | 100 [48 to 100]

2. Secondary Outcome: Change in Ocular Quantitative Myasthenia Score From Baseline to Week 16
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | -2.25 [-5.56 to 1.05] | -0.05 [-3.71 to 3.60]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; Mean Ocular QMG Changes from Baseline to Week 16 . 95% CI and p-values obtained from the analysis of covariance model to adjust for the baseline value of the outcome variable; Test type: Non-Inferiority or Equivalence — N=80, (40 per group), 80% power to detect a group difference of 30%-35% and 5% significance level; p = 0.37, ANCOVA; ANCOVA used to compare mean values adjusting for the baseline value; Mean Difference (Final Values) = -2.20, 95% CI 2-sided [-7.20 to 2.8] — QMG Score ranges from 0-15, where 0 is normal and a reduction in score represents imrovement

3. Secondary Outcome: Change in Quality of Life as Measured by the NEI-VFQ-25 Measures
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | 10.7 [4.75 to 16.64] | 4.14 [-2.54 to 10.82]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; Mean Change in quality of life as measured by the NEI-VFQ-25 at the end of Double- Blinded Treatment. 95% CI and p-values obtained from the analysis of covariance model to adjust for the baseline value of the outcome variable; Test type: Non-Inferiority or Equivalence — Mean Change in quality of life as measured by the NEI-VFQ-25 at the end of Double- Blinded Treatment; p = 0.13, ANCOVA; Mean Difference (Net) = 6.56, 95% CI 2-sided [-2.59 to 15.71] — Scores ranges fro 0-100 , where 100 is normal and an increase in score represents an improvement

4. Secondary Outcome: Change in Quality of Life as Measured by the MG-QOL-15 Score
Time Frame: 4 Months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | -6.3 [-10.11 to -2.50] | -2.5 [-6.30 to 1.31]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; Mean Change in quality if life as measured by the MG-QOL-15 score at the end of Double- Blinded Treatment. 95% CI and p-values obtained from the analysis of covariance model to adjust for the baseline value of the outcome variable; Test type: Non-Inferiority or Equivalence — Mean Change in quality if life as measured by the MG-QOL-15 score at the end of Double- Blinded Treatment; p = 0.15, ANCOVA; Mean Difference (Final Values) = -3.81, 95% CI 2-sided [-9.37 to 1.75] — Ranges from 0-60, where 0 is Normal and a reduction in score represents improvement

5. Secondary Outcome: Change in Quality of Life as Measured by the 10-Item Neuro-ophthalmological Supplement to the NEI-VFQ-25
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | 15.28 [-0.62 to 31.17] | -1.7 [-19.83 to 16.43]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; Mean Change NEI-VFQ-25 10 item neuro-opthtalmological supplement score baseline to week 16. 95% CI and p-values obtained from the analysis of covariance model to adjust for the baseline value of the outcome variable; Test type: Non-Inferiority or Equivalence — Mean Change NEI-VFQ-25 10 item neuro-opthtalmological supplement score baseline to week 16; p = 0.16, ANCOVA; Mean Difference (Final Values) = 16.98, 95% CI 2-sided [-9.22 to 43.17] — Ranges 0-100, where 100 is normal and an increase in score represents an improvement

ADVERSE EVENTS:
Time Frame: Adverse Events After Randomization
Arm/Group | Prednisone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone (N=6) | Placebo (N=5)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
DIVERTICULAR ABCESS (Infections and infestations) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
GI BLEED (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone (N=6) | Placebo (N=5)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 2 (2) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
INSOMNIA (Nervous system disorders) | 0 (0) | 1 (1)
AGITATION (Nervous system disorders) | 1 (1) | 0 (0)
ANXIETY (Nervous system disorders) | 0 (0) | 1 (1)
ARRHYTMIA (Cardiac disorders) | 1 (1) | 0 (0)
BLEPHAROSPASM (Nervous system disorders) | 1 (1) | 0 (0)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONDUCTION DISORDER (Cardiac disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
EDEMA: HEAD AND NECK (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
FACE FASCICULATION (RIGHT SIDE) (Nervous system disorders) | 1 (1) | 0 (0)
HEMATOMA (Vascular disorders) | 1 (1) | 0 (0)
IMPAIRED GLUCOSE TOLERANCE (Endocrine disorders) | 1 (1) | 0 (0)
EYE PAIN(POCKET IN EYE) (Eye disorders) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
EYE FASCICULLATION (Nervous system disorders) | 1 (1) | 0 (0)
WEIGHT GAIN (Endocrine disorders) | 2 (2) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BLURRED VISION (Nervous system disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No